CLINICAL TRIAL: NCT00758927
Title: The Effects of OMACOR on the LDL Sub-fraction in Korean Type 2 Diabetic Patients With Combined Hyperlipidemia
Brief Title: The Effects of Omega-3 Fatty Acid (OMACOR) on the Low-density Lipoprotein (LDL) Sub-fraction in Type 2 Diabetic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inje University (Other)
Collaborators: Kuhnil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Jeong Hyun Park/Professor, Pusan Paik Hospital, Inje University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-OM-9408
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Diabetes Mellitus, Type 2; Hypercholesterolemia; Hypertriglyceridemia
Keywords: diabetes mellitus; combined hyperlipidemia; OMACOR; small dense LDL; HDL subfraction
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypercholesterolemia; Hypertriglyceridemia; Diabetes Mellitus | interventions — Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): Placebo administration for 10 weeks with exercise and diet therapy
  Interventions: Drug: Placebo control
- 1 (Experimental): Omacor 4 gram per day with exercise and diet therapy for 10 weeks
  Interventions: Drug: Omega-3 acid 4 grams per day

INTERVENTIONS:
Drug: Omega-3 acid 4 grams per day — OMACOR 4 grams per day is administered simultaneously with exercise and diet therapy
  Other Names: OMACOR
  Arms: 1
Drug: Placebo control — Placebo will be administered simultaneously with exercise and diet therapy in same intensity with the experimental arm
  Other Names: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to verify the possible effects of OMACOR(omega-3 fatty acid) on the percentage change of small dense LDL fraction in type 2 diabetic patients with combined hyperlipidemia, we perform open-label prospective randomized multi-institutional phase IV study.

DETAILED DESCRIPTION:
The main cause of mortality in type 2 diabetes mellitus is a cardiovascular disease. Among the many risk factors of atherosclerosis in diabetic patients, LDL(low density lipoprotein) cholesterol is now being regarded as one of the most important modifiable one. Recent researches have revealed that the plasma LDL could be sub-divided according to the size of the particles into large buoyant LDL and small dense LDL. Small dense LDL is very atherogenic. Increased plasma triglyceride and the presence of insulin resistance are proved to be positively correlated well with the amount of small dense LDL in diabetic patients.

We would like to see omega-3 acid(OMACOR) which is now widely used in clinical practice to decrease plasma triglyceride could change the amount of plasma small dense LDL in type 2 diabetic patients with combined hyperlipidemia.

This trial is consisted of 6 weeks of wash out for the patients already taking statin. After that, daily 4 grams of omega-3 acid(OMACOR) will be administered for 10 weeks. Before and after the administration of study drug, we will measure the change of the amount of plasma small dense LDL via ultracentrifuge/non-denaturing polyacrylamide gel electrophoresis followed by oil red O and coomassie blue staining. As a secondary outcome measure, we will also assess the change of HDL(high density lipoprotein) cholesterol sub-type by the same method.

ELIGIBILITY:
Inclusion Criteria:

* Agreed for informed consent
* Age between 40-70 years old
* Type 2 diabetes mellitus
* Combined hyperlipidemia
* Serum triglyceride level between 200-500(mg/dl)
* No sudden change of glucose lowering therapies during trial, anticipated

Exclusion Criteria:

* Hypersensitivity to OMACOR(Omega-3 fatty acid)
* Alcoholics
* Pregnancy
* Proliferative diabetic retinopathy
* Patients already taking fibrates
* Enrolled in other clinical trials during the recent 3 months
* Severe ischemic heart disease, liver disease, neurological disease
* AST/ALT level 2 folds above the normal reference level
* Psychiatric disorder not adequately controlled
* Serum creatinine over 2.0 (mg/dl)
* Previous pancreatic surgery
* Patients who can not maintain regular diet

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-04 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Percentage change of plasma small dense LDL measured by ultracentrifuge-non denaturing polyacrylamide gel electrophoresis | April 2009

SECONDARY OUTCOMES:
The percentage change of plasma HDL sub-fraction measured by ultracentrifuge-non denaturing polyacrylamide gel electrophoresis | April 2009

CONTACTS AND LOCATIONS:
Overall Officials: Jeong H Park, M.D., Ph.D., Principal Investigator — Director, Paik Diabetes Center, Pusan Paik Hospital, Inje University
Locations (3):
- South Korea (3):
  - Dong-A University Medical Center, Busan
  - Paik Diabetes Center, Busan
  - Endocrinology and Metabolism, Maryknoll General Hospital, Busan